CLINICAL TRIAL: NCT05384444
Title: Effect of Perioperative Dietary Restriction Strategy on Postoperative Recovery and Outcomes of Patients With Colorectal Cancer : a Multicenter Prospective, Randomized, Controlled Study
Brief Title: Effect of FMD on Colorectal Cancer Patients
Acronym: FCRC22
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Cancer Hospital, China (Other); Huashan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tongji Hospital (Other); Changhai Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Changhong Miao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-063(2)
Record Dates: First submitted 2022-04-13; First posted 2022-05-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Fasting Mimicking Diet; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Concealed allocation: the statisticians formulate the randomization scheme and generates the random number.
Masking Description: Allocation concealment：an independent researcher implements the randomized allocation scheme to ensure that the subjects and the researchers who screen the subjects are unable to know the subsequent subjects in advance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting mimicking diet (Experimental): The cyclic FMD diet consists of a 5 day regimen: day 1 diet of the diet supplies ~1000 kcal (10% protein, 56% fat, 34% carbohydrate), day 2-5 are identical in formulation and provide 800 kcal (9% protein, 44% fat, 47% carbohydrate). At least 4 cyclic FMDs will be performed after operation.
  Interventions: Other: Fasting mimicking diet
- regular diet (No Intervention): regular diet

INTERVENTIONS:
Other: Fasting mimicking diet — The fasting mimicking diet consists of a 5 day regimen: day 1 diet of the diet supplies ~1000 kcal (10% protein, 56% fat, 34% carbohydrate), day 2-5 are identical in formulation and provide 800 kcal (9% protein, 44% fat, 47% carbohydrate). At least 4 cyclic FMDs will be performed after operation.
  Arms: Fasting mimicking diet

SUMMARY:
Extensive preclinical evidence suggests that short-term fasting and fasting mimicking diets (FMDs) can protect healthy cells and render cancer cells more vulnerable to chemotherapy and other therapies. However, fasting is difficult for the old and frail subjects.Therefore, FMDs may be more suitable for postoperative dietary intervention in cancer patients. Colorectal tumors have high glucose consumption, which makes tumor cells very sensitive to changes in nutritional metabolism of the surrounding environment (such as diet restriction / fasting). Previous studies have shown that cyclic FMDs are safe and feasible for cancer patients receiving chemotherapy alone. However, the effects of the FMD in patients under radical surgery for colorectal cancer have not been evaluated so far. This study aims to evaluate the impact of FMDs on postoperative recovery and outcomes of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 80 years old
2. Patients undergoing radical colorectal cancer resection for the first time
3. Preoperative clinical tumor stage III
4. ASA grade I-III grade
5. With BMI 19-32 kg/m2
6. Adequate liver function, adequate renal function and normal cardiac function
7. Willing to participate in the research of the subject and agree to follow up regularly

Exclusion Criteria:

1. Evidence of distant metastasis before surgery
2. Before surgery, have received treatment of neoadjuvant chemotherapy
3. Type 1 diabetes or intensive insulin therapy
4. Allergies for FMD content
5. Combined with severe primary diseases such as severe immune system or autoimmune system or long-term using of glucocorticoids or immunosuppressant
6. History of opioid abuse, mental illness or cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 3 years
  DFS is defined as the interval between the date of first treatment and the date of recurrence or metastasis or secondary primary tumor or death.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  OS is defined as the interval between the date of first treatment and the date of death due to any reason.
Weight, height and BMI | 3 years
  Weight in kilograms, height in meters, weight and height will be combined to report BMI in kg/m^2
upper arm circumference and waistline | 3 years
  upper arm circumference and waistline in centimeters
heart rate, blood pressure and basal metabolic rate | 3 years
  heart rate in bpm and blood pressure in mmHg, heart rate and blood pressure will be combined to report basal metabolic rate
body composition | after randomization, before discharge, before and at the completion of each FMD cycle.
  Body composition (fat-free mass, fat mass, phase angle, extracellular mass-to-body cell mass ratio (ECM/BCM), total body water and intracellular water, bioelectrical impedance) measurements are analyzed with a Single Frequency Bioimpedance Analyzer (Inbody 770, South Korea).
plasma protein | 3 years
  plasma protein will be recorded before and at the completion of each FMD cycle.
Nutritional status | 3 years
  Patient-Generated Subjective Global Assessment (PG-SGA) to measure nutritional status. Higher scores (0-53 scale) indicate a worse nutritional status.
Feasibility of the FMD in colorectal cancer patients | 3 years
  Feasibility is defined as the ability of the patient to comply with the prescribed dietary regimen. It will be assessed through the analysis of food diaries filled by patients during the five days of each FMD cycle.
Quality of life(QOL) | 3 years
  QOL is respectively evaluated by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30). Higher scores (0-100 scale) on the functional scales indicate a better QoL.
Exercise tolerance | 3 years
  Metabolic Equivalents (METs) scale to measure exercise tolerance. Higher scores (1-10 scale) indicate a better exercise tolerance.
Postoperative pain | 3 years
  Numerical Rating Scale (NRS) to evaluate pain degree. Higher scores (0-10 scale) indicate a more severe pain.
Occurrence of clinical complications | 3 years
  Any postoperative complications will be recorded.
Neutrophil to Lymphocyte Ratio (NLR) | 3 years
  NLR will be measured after randomization, before discharge and before and at the completion of each FMD cycle.
Lymphocyte to Monocyte Ratio (LMR) | 3 years
  LMR will be measured after randomization, before discharge and before and at the completion of each FMD cycle.
Systemic immune-inflammation index (SII) | 3 years
  SII will be measured after randomization, before discharge and before and at the completion of each FMD cycle.
Inflammatory factor level | 3 years
  IL-1β,IL-2,IL-4,IL-5,IL-6,IL-8,IL-10,IL-17A,IL-17F,TNF-α，TNF-β in pg/ml
T Lymphocyte cell count | 3 years
  T lymphocyte cell count before and at the completion of each FMD cycle.
insulin-like growth factor-I (IGF-I) | 3years
  Insulin-like growth factor-I (IGF-I) in ng/ml. IGF-I will be measured before and at the completion of each FMD cycle.
Glucose | 3years
  Glucose in mmol/L. Glucose will be measured before and at the completion of each FMD cycle.
insulin | 3years
  Insulin in U/L. Insulin will be measured before and at the completion of each FMD cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Miaomiao Guo, Dr, Principal Investigator — Shanghai Zhongshan Hospital; Meilin Weng, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (6):
- China (6):
  - Fudan University Huashan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality
  - Fudan University,ZhongShan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Naval Medical University,, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital,Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital,Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No